CLINICAL TRIAL: NCT03202732
Title: DiabetesFlex - Patient Involvement and Patient-reported Outcome Measures in Type 1 Diabetes: A Randomised Controlled Trial and Interview Study
Brief Title: DiabetesFlex - Patient Involvement and Patient-reported Outcome Measures in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Annesofie Lunde Jensen (Other)
Responsible Party: Sponsor-Investigator, Annesofie Lunde Jensen, Clinical nursespecialist postdoc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DiabetesFlex2017
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Self-management; Patient Activeted measure; Patient-reported outcome; Type 1 diabetes Mellitus; Non-inferiority study
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DiabetesFlex (Other): In DiabetesFlex intervention, patients are offered 3 consultations/year. One mandatory consultations (30 minutes). The patient, an endocrinologist and a diabetes nurse attend.
  Two optional consultations, patients can choose between face-to-face consultations, a telephone consultation or to cancel the consultation.
  Ahead of the consultations, patients fill out the AmbuFlex Diabetes questionnaire and deliver a blood and urine sample.
  Based on the patient's response to the AmbuFlex Diabetes questionnaire, the result of the blood sample and the urine sample, the diabetes nurse assign the patient to a face-to-face consultation, a telephone consultation or no consultation with an endocrinologist, a diabetes nurse or a dietician.
  Interventions: Other: DiabetesFlex
- Standard care (No Intervention): Standard diabetes care consists of 3 consultations (15 minutes)/year with a physician or a diabetes nurse by turns.
  Ahead of the consultation patients send in a blood sample for measuring HgA1c, urine sample for measuring urin-albumin creatinin ratio and other blood samples depending of arrangements made in the last consultation.
  Once a year in relation to a consultation, patients fill in the Problem Area In Diabetes (PAID) (20) scale together. Furthermore, based on the patients or healthcare professional judgement, patients see a dietician when needed.

INTERVENTIONS:
Other: DiabetesFlex — DiabetesFlex consist of one mandatory and two optional consultations. Before the consultations patients receive the AmbuFlex Diabetes questionnaire.
  The AmbuFlex Diabetes questionnaire is based on both validated questionnaires and clinical consensus. The AmbuFlex Diabetes questionnaire consists of: SF36 well-being question, WHO-5 Well-being Index. Questions concerning: HgA1c, home-based blood pressure monitoring, incidents of hypoglycemia, diabetes complications, regular eye check, regular food check, erectile dysfunction and peripheral neuropathy, The PAID scale, Topics patients may want to talk with the health care professional about, the patient's evaluation of the need for diabetes care. View the AmbuFlex Diabetes questionnaire at the homepage: www.diabetesflex.auh.dk.
  Arms: DiabetesFlex

SUMMARY:
The aim of this study is to investigate the effect of the use of DiabetesFlex in diabetes care compared to standard care in relation to patient involvement and relevance for specific group of persons with T1DM.

The investigators hypothesize that the use of DiabetesFlex will lead to a higher degree of patient in-volvement, improved glycaemic control and a decrease in total number of consultations compared to standard care. Furthermore, the investigators aim to identify if a specific sub-population within the T1DM population will benefit significantly from the intervention.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic condition, and provision of individual and effective diabetes care is a major challenge. The is a lack of evidence on the optimal frequency of attending outpatient clinics for persons with T1DM.

The use of patient-reported outcome (PRO) measures in diabetes care area are limited and none existing in a Danish context. This includes studies, which combine PRO measure with diabetes management, patient involvement and self-management.

The study will generate knowledge and directions for ways to reframe and to optimize the future management of diabetes care.

ELIGIBILITY:
Inclusion Criteria:

Age over 18 years Have had T1DM for more than 1 years Be able to use the Danish-language general website on healthcare www.sundhed.dk Be mentally well functioning Understand and read Danish Access to internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
HbA1c | 15 mounth
  Non-inferiority with respect to HbA1c

SECONDARY OUTCOMES:
General health will be assessed by items from the SF-36 questionnaire | 15 mounth
  General health will be measured at baseline and after 15 mounth
Health literacy will be assessed by The Health Literacy Questionnaire (sub scale 6 and 9) | 15 mounth
  Health literacy will be measured at baseline and after 15 months.
Well-being will be assessed by the WHO-5 Well-being Index | 15 mounth
  Well-being will be measured at baseline and after 15 months.
Patient Activated Measure (PAM) | 15 mounth
  Patient Activated Measure (PAM) will be measured at baseline and after 15 months.
"Generic questions concerning patient involvement" is validate by "DEFACTUM" | 15 mounth
  Patient involvement will be measured at baseline and after 15 months.
The problem Areas In Diabetes Scale (PAID) | 15 mounth
  PAID will be measured at baseline and after 15 months.
Blood pressure | 15 mounth
  Blood pressure will be measured at baseline and after 15 months.
Urine albumine/creatinine ratio | 15 mounth
  urine albumine/creatinine ratio will be measured at baseline and after 15 months.
Number and type consultations | 15 mounth
  Consultations consists of face-to-face, telephone, cancel, registered non-attendance and health care professional involved in the consultation will be measured after 15 mounth
Mortality | 15 mounth
  Mortality will be measured after 15 months.

CONTACTS AND LOCATIONS:
Overall Officials: Annesofie L. Jensen, Postdoc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aahurs University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No